CLINICAL TRIAL: NCT01215435
Title: An Open Labelled, Randomised, Parallel Trial; Efficacy and Safety Comparison of Two Different Biphasic Insulin Aspart 30 Treatment Initiation Regimens Followed by Intensification in Subjects With Type 2 Diabetes Mellitus Not Achieving Glycaemic Targets on OADs Alone in Iran
Brief Title: Comparison of Two Biphasic Insulin Aspart 30 Treatment Regimens in Subjects With Type 2 Diabetes Not Achieving HbA1c Treatment Targets on OADs Alone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIASP-3858; U1111-1116-2121 (Other: WHO)
Record Dates: First submitted 2010-10-01; First posted 2010-10-06 (Estimated); Results first posted 2013-11-25 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-breakfast BIAsp 30 (Experimental)
  Interventions: Drug: biphasic insulin aspart 30
- Pre-dinner BIAsp 30 (Experimental)
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — Administered subcutaneously (under the skin) once daily, before breakfast. The trial has 3 treatment phases for both treatment arms
  Arms: Pre-breakfast BIAsp 30
Drug: biphasic insulin aspart 30 — Administered subcutaneously (under the skin) once daily, before dinner. The trial has 3 treatment phases for both treatment arms
  Arms: Pre-dinner BIAsp 30

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to compare the glycaemic control when subjects initiate a biphasic insulin aspart 30 treatment followed by an intensified treatment if treatment target of HbA1c below 7% is not reached by OAD (oral anti-diabetic drugs) alone.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes for a minimum of 6 months prior to Visit 1
* HbA1c at least 7.0 % - maximum 11 % at screening
* Subject is insulin naïve (short-term insulin treatment of up to 14 days is allowed)
* An antidiabetic regimen that has been stable for at least 3 months prior to screening
* An antidiabetic regimen that includes a minimum of 2 OADs
* OADs dosed at least 50% of the maximum recommended dose

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product(s) or related products
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptive measures as required by local law or practice)
* The receipt of any investigational medicinal product within one month prior to this trial
* Suffer from a life threatening disease (cancer)
* Cardiac disease: class III or IV congestive heart failure (CHF), unstable angina, and or any myocardial infarction (treated or untreated) within 6 months prior to screening
* Hepatic insufficiency (Alanine aminotransferase (ALT) or Aspartate aminotransferase (AST) above 2 times the central laboratory's upper reference limit)
* Renal insufficiency (serum creatinine above 1.6 mg/dl for males; 1.4 mg/dl for females
* Recurrent hypoglycaemia or hypoglycaemic unawareness
* Anemia (haemoglobin below 10 mg/dl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2011-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Tehran, Iran

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 5 sites in Iran
Pre-assignment Details: Subjects were on a stable antidiabetic regimen which includes a minimum of 2 OADs, daily for at least 3 months prior to screening. OAD doses were at least 50 percent of the maximum recommended dose.
Groups:
- Pre-breakfast BIAsp 30: Subjects were started on BIAsp 30 (a biphasic formulation of insulin aspart (IAsp) in which 30% is soluble and the remaining 70% is protaminized insulin aspart) subcutaneously once daily (OD) pre-breakfast. Then they were intensified to twice daily (BID) or thrice daily (TID) if glycaemic control is not achieved, within three 12 weeks of treatment phases by titrating according to SMBG levels.
- Pre-dinner BIAsp 30: Subjects were started on BIAsp 30 (a biphasic formulation of insulin aspart (IAsp) in which 30% is soluble and the remaining 70% is protaminized insulin aspart) subcutaneously once daily (OD) pre-dinner. Then they were intensified to BID or TID if glycaemic control is not achieved, within three 12 weeks of treatment phases by titrating according to SMBG levels.
Period: Overall Study
Arm/Group | Pre-breakfast BIAsp 30 | Pre-dinner BIAsp 30
Started | 122 | 123
Completed | 103 | 107
Not Completed | 19 | 16
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal Criteria | 8 | 11
Not completed — Lost to Follow-up | 3 | 0
Not completed — Unclassified | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-breakfast BIAsp 30 | Pre-dinner BIAsp 30 | Total
Number analyzed (Participants) | 122 | 123 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (9.32) | 54.8 (10.32) | 55.2 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 74 | 146
  Male | 50 | 49 | 99
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 9.1 (1.07) | 9.2 (1.00) | 9.2 (1.04)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 192.7 (68.56) | 199.3 (63.80) | 196.0 (66.16)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c) From Baseline to Week 11
Description: Estimated mean change from baseline in HbA1c after 11 weeks of treatment
Time Frame: Week 0, Week 11
Population: Full analysis set (FAS) includes all randomised subjects and missing data was imputed using baseline observation carried forward (BOCF)
Measure: Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | Pre-breakfast BIAsp 30 | Pre-dinner BIAsp 30
Number analyzed (Participants) | 122 | 123
percentage of glycosylated haemoglobin | -1.04 (0.10) | -0.90 (0.10)
Statistical Analysis 1: Comparison: Pre-breakfast BIAsp 30 vs Pre-dinner BIAsp 30; H0: D > 0.4% against H1: D ≤ 0.4% where D is the mean treatment difference for change in HbA1c (pre-breakfast OD minus pre-dinner OD); Test type: Non-Inferiority or Equivalence — Non-inferiority was considered confirmed if the upper bound of the two-sided 95% confidence interval for the mean HbA1c treatment difference was below or equal to 0.4%. This is equivalent to using a one-sided test of size 2.5%; p < 0.001, Regression, Linear; Estimated treatment difference, Mean = -0.14, 95% CI [-0.40 to 0.13]

2. Secondary Outcome: Change in FPG (Fasting Plasma Glucose) From Baseline to Week 36
Description: Estimated mean change from baseline in FPG after 36 weeks of treatment
Time Frame: Week 0, Week 36
Population: Full analysis set (FAS) includes all randomised subjects and missing data was imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Pre-breakfast BIAsp 30 | Pre-dinner BIAsp 30
Number analyzed (Participants) | 122 | 123
mg/dL | -61.57 (4.50) | -58.43 (4.48)
Statistical Analysis 1: Comparison: Pre-breakfast BIAsp 30 vs Pre-dinner BIAsp 30; Test type: Superiority or Other; p = 0.6215, Regression, Linear; Estimated treatment difference, Mean = -3.14, 95% CI [-15.65 to 9.37]

3. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes
Description: A hypoglycaemic episode will be defined as treatment emergent if the onset of the episode is on or after the first day of trial product, and no later than the last day on trial product.
Time Frame: Week 0 to Week 36
Population: Safety analysis set includes all subjects who received at least one dose of the trial product.
Measure: Number; unit: episodes
Arm/Group | Pre-breakfast BIAsp 30 | Pre-dinner BIAsp 30
Number analyzed (Participants) | 122 | 123
episodes | 1181 | 953

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a timeframe of 36 weeks +14 days follow-up.
Description: Safety analysis set includes all subjects who received at least one dose of the trial product.
Arm/Group | Pre-breakfast BIAsp 30 | Pre-dinner BIAsp 30
Serious Adverse Events (participants affected / at risk) | 3/122 | 4/123
Other Adverse Events (participants affected / at risk) | 16/122 | 19/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-breakfast BIAsp 30 (N=122) | Pre-dinner BIAsp 30 (N=123)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-breakfast BIAsp 30 (N=122) | Pre-dinner BIAsp 30 (N=123)
Nasopharyngitis (Infections and infestations) | 7 (8) | 8 (13)
Hyperlipidaemia (Metabolism and nutrition disorders) | 9 (9) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol.